CLINICAL TRIAL: NCT02959229
Title: Systematic Randomized , Single Blinded, Placebo-Controlled Trial of Early Versus Late Lactoferrin in Prevention of Neonatal Sepsis
Brief Title: Early Versus Late Lactoferrin in Prevention of Neonatal Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Atef Nagy Mohamed, clinical researcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU M.S 23/2016
Record Dates: First submitted 2016-10-27; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Neonatal Sepsis
Keywords: Late onset sepsis; Bovine Lactoferrin
MeSH Terms: conditions — Neonatal Sepsis | interventions — Lactoferrin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Early Lactoferrin Group (Experimental): Oral Bovine Lactoferrin 100 mg/day once starting on day 1 of life and continued for 4-6 weeks.
  Interventions: Drug: Lactoferrin
- Late Lactoferrin Group (Experimental): Oral Bovine Lactoferrin 100 mg/day once starting on day 3 of life and continued for 4-6 weeks.
  Interventions: Drug: Lactoferrin
- Placebo Group (Active Comparator): placebo in form of distilled water once starting on day 1 of life and continued for 4-6 weeks.
  Interventions: Drug: Placebo (for Lactoferrin)

INTERVENTIONS:
Drug: Lactoferrin
  Other Names: Bovine Lactoferrin
  Arms: Early Lactoferrin Group; Late Lactoferrin Group
Drug: Placebo (for Lactoferrin) — placebo in form of distilled water
  Arms: Placebo Group

SUMMARY:
The present study was designed to evaluate the effectiveness of oral lactoferrin in prevention of neonatal sepsis with comparison early (1st day) versus late (48-72 hours) Lactoferrin administration, Secondary aim was to study effect of Lactoferrin administration on serum Ferritin and follow up long term outcome (Bronchopulmonary dysplasia, retinopathy of prematurity and necrotizing enterocolitis.

DETAILED DESCRIPTION:
This study was carried out on 180 preterm neonates(< 37 weeks of gestation counting from the first day of the Last Menstrual Period and confirmed by Ballard score) admitted to the Neonatal Intensive Care Units of Ain Shams University Hospitals in the period from August 2014 to December 2015.

Enrolled subjects were further randomly subdivided into three groups according to the dose regimen of Lactoferrin supplementation.

* Group A: (60 preterm neonates) who received oral Lactoferrin supplementation in a dose of 100 mg/day starting on day 1 and continue for 4-6 weeks.
* Group B: (60 preterm neonates) who received oral Lactoferrin supplementation in a dose of 100 mg/day starting on day 3 (48hrs-72hrs) of life and continue for 4-6 weeks.
* Group C: (60 preterm neonates) who match the subjected neonates, received placebo in form of distilled water.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with a < 37 weeks of gestation counting from the first day of the Last Menstrual Period.
2. Preterm neonates are breast fed, artificially fed or on total parenteral nutrition.
3. Preterm neonates born in, or referred to our Neonatal Intensive Care Unit in the first day of life free from infection and not fed.

Exclusion Criteria:

1. Neonates with underlying gastrointestinal problems that prevent oral intake.
2. Neonates with predisposing conditions that profoundly affect growth and development (chromosomal abnormalities, structural brain anomalies, severe congenital abnormalities).
3. Neonates with a family background of cow milk allergy.
4. Neonates who will not have the chance to complete the study time (who will be referred to another hospitals).
5. Neonates with early onset sepsis.
6. Neonates whose parents decline to participate.

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of oral Lactoferrin in prevention of neonatal sepsis according to Tollner score, hematological scoring system (HSS) and positive blood culture. | 4-6 weeks of life
Compare early (1st day) versus late (48-72 hours) Lactoferrin administration on neonatal sepsis according to Tollner score, hematological scoring system (HSS) and positive blood culture | 4-6 weeks of life

SECONDARY OUTCOMES:
Effect of Lactoferrin supplementation on long term complications | 4-6 weeks of life
  Long term complications as:
  Broncho-Pulmonary Dysplasia using clinical symptoms and signs and chest X ray findings.
  Retinopathy of Prematurity using the International Classification of Retinopathy of Prematurity (ICROP).
  Necrotizing Enterocolitis using Modified Bell's criteria for staging Necrotizing Enterocolitis.
any reported side effects for Bovine Lactoferrin | 4-6 weeks of life

CONTACTS AND LOCATIONS:
Overall Officials: Ghada I Ghad, Professor, Study Director — Ain Shams University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaur G, Gathwala G. Efficacy of Bovine Lactoferrin Supplementation in Preventing Late-onset Sepsis in low Birth Weight Neonates: A Randomized Placebo-Controlled Clinical Trial. J Trop Pediatr. 2015 Oct;61(5):370-6. doi: 10.1093/tropej/fmv044. Epub 2015 Jul 29. PMID 26224129
- [Background] Manzoni P, Meyer M, Stolfi I, Rinaldi M, Cattani S, Pugni L, Romeo MG, Messner H, Decembrino L, Laforgia N, Vagnarelli F, Memo L, Bordignon L, Maule M, Gallo E, Mostert M, Quercia M, Bollani L, Pedicino R, Renzullo L, Betta P, Ferrari F, Alexander T, Magaldi R, Farina D, Mosca F, Stronati M. Bovine lactoferrin supplementation for prevention of necrotizing enterocolitis in very-low-birth-weight neonates: a randomized clinical trial. Early Hum Dev. 2014 Mar;90 Suppl 1:S60-5. doi: 10.1016/S0378-3782(14)70020-9. PMID 24709463